CLINICAL TRIAL: NCT06355245
Title: MEDECA - Markers in Early Detection of Cancer
Acronym: MEDECA
Status: Recruiting | Type: Observational
Sponsor: Danderyd Hospital (Other)
Responsible Party: Principal Investigator, Charlotte Thålin, M.D., Ph.D. Senior consultant in internal medicine, Danderyd Hospital
Other Study IDs: 2017/2160-31/1
Record Dates: First submitted 2024-01-10; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Cancer; Diagnosis
MeSH Terms: conditions — Neoplasms; Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with unspecific symptoms: Patients referred to the Diagnostic Center at Danderyd Hospital (DC DS), a multidisciplinary diagnostic center referral pathway for patients with radiological findings suggestive of metastasis without known primary tumor or suspicion of serious but unspecific symptoms.
  Interventions: Diagnostic Test: Blood sampling

INTERVENTIONS:
Diagnostic Test: Blood sampling — Collection of blood samples

SUMMARY:
Early diagnosis of cancer is key for improving patient outcomes, but cancers are difficult to diagnose if patients present with unspecific symptoms. The principal objective of the MEDECA (Markers in Early Detection of Cancer) study is to identify a multi-analyte blood test that can detect and map occult cancer within a mixed population of patients presenting with serious but unspecific symptoms. The study will include 1500 patients referred to the Diagnostic Center at Danderyd Hospital (DC DS), a multidisciplinary diagnostic center referral pathway for patients with radiological findings suggestive of metastasis without known primary tumor or suspicion of serious but unspecific symptoms. Blood samples are collected prior to a standardized and extensive cancer diagnostic work-up, including an expanded panel of biochemical analyses and extensive imaging such as computed tomography or magnetic resonance investigations. In collaboration with world-leading international scientists, the blood samples will be analyzed for a panel of novel and established blood biomarkers predictive of an underlying cancer, including markers of neutrophil extracellular traps, circulating tumor DNA, platelet mRNA profiling, affinity-based proteomics and nuclear magnetic resonance metabolomics. The diagnostic accuracy of the blood biomarkers with respect to cancer detection during the diagnostic work-up will be analyzed through machine learning.

ELIGIBILITY:
Inclusion Criteria:

- Age above 18 years

One or more of the following symptoms/clinical signs:

* General malaise
* Severe tiredness
* Unintentional weight loss
* Fever of unknown cause
* Uncharacteristic pain for >4 weeks
* Abnormal laboratory tests (e.g., anemia, elevated alkaline phosphatase levels, erythrocyte sedimentation rate (ESR), calcium etc.)
* Diffuse pain without explanation
* Marked increase in drug usage
* Increasing health service seeking behavior
* Radiological findings suggestive of metastasis without known primary tumor or suspicion

Exclusion Criteria:

* Unwillingness to participate in the study
* Age below 18 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study participants are enrolled at the first visit to DC DS. The criteria for referral to DC DS are radiological findings suggestive of metastasis without known primary tumor or suspicion of serious illness based on one or more of the following symptoms: general malaise, severe tiredness, unintentional weight loss, fever of unknown cause, uncharacteristic pain for >4 weeks, abnormal laboratory tests (e.g., anemia, elevated alkaline phosphatase levels, erythrocyte sedimentation rate (ESR), calcium etc.), diffuse pain, marked increase in drug usage or increasing health service seeking behavior.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Cancer diagnosis | During diagnostic work-up (within six months)
  Patients undergo an extensive diagnostic work-up and diagnoses are obtained from medical records

SECONDARY OUTCOMES:
Other diagnosis | During the diagnostic work-up (within six months) as well as in a one-year follow-up
  Patients undergo an extensive diagnostic work-up and diagnoses are obtained from medical records
Mortality | Within 1 year from inclusion
  Will be obtained from medical records
Cancer diagnosis | Within 1 year from inclusion
  Will be obtained from medical records

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Thålin, M.D., Ph.D, Principal Investigator — Danderyd Hospital Karolinska Institutet
Locations (1):
- Danderyd Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No